CLINICAL TRIAL: NCT04796441
Title: Clinical Study of Universal CAR-γδT Cell Injection in the Treatment of Patients With Relapsed AML After Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hebei Senlang Biotechnology Inc., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAR-γδT cell for AML
Record Dates: First submitted 2021-03-08; First posted 2021-03-12 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: AML
Keywords: AML γδT CAR-

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR--γδT (Experimental): Patients will be treated with CAR--γδT cells
  Interventions: Biological: CAR-γδT

INTERVENTIONS:
Biological: CAR-γδT — Biological: CAR-γδT; Drug: Cyclophosphamide,Fludarabine; Procedure: Leukapheresis;
  Other Names: CD19 CAR-T

SUMMARY:
This is an open single-arm clinical study aimed at evaluating the efficacy and safety of universal γδT cell injection in the treatment of patients with relapsed AML after transplantation

DETAILED DESCRIPTION:
Main purpose: To evaluate the safety and effectiveness of universal CAR-γδT cell injection in the treatment of patients with relapsed AML after transplantation

Secondary purpose: to investigate the in vivo dynamics characteristics of universal CAR-γδT cells after infusion and explore reasonable therapeutic doses through climbing tests in different dose groups.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with clinically diagnosed recurrence of AML after receiving transplant therapy;
2. Flow cytometry (FCM) or immunohistochemical detection of tumor cells confirmed CD123 positive;
3. Age ≥2 years old and <65 years old;
4. Survival is expected to be greater than 3 months from the date of signing of the informed consent;
5. KPS 80 points or more;
6. The functions of vital organs shall meet the following conditions:

1) EF>50%, and no obvious ECG abnormality; 2) SpO2 90% or more; 3) Cr 2.5 ULN or less; 4) ALT And AST≤5ULN, TBil≤3ULN; 7. Subjects who plan to become pregnant must agree before study enrollment and after study duration of 6 months Use contraception; Inform the investigator immediately if the subject is pregnant or suspected to be pregnant; 8. Subject or guardian understands and signs the informed consent;

Exclusion Criteria:

* 1. Other diseases that have not been effectively controlled, including but not limited to persistent or poorly controlled infections and diseases Congestive heart failure, unstable angina pectoris, arrhythmias, poorly controlled lung disease Or mental illness; 2. Other active malignant tumors; 3. Complicated with severe infection that cannot be effectively controlled; 4. Active hepatitis B (HBVDNA) or HCV RNA [HCVRNA] test was positive); 5. Human immunodeficiency virus (HIV) infection or syphilis infection; 6. Have a history of severe allergy to biological products (including antibiotics); 7. Acute graft-versus-host reaction (GVHD) was still present one month after discontinuation of immunosuppressant therapy Allogeneic hematopoietic stem cell transplantation patients; 8. Female subjects are in pregnancy and lactation; 9. Active autoimmune diseases requiring systemic immunosuppression; 10. Conditions that the investigator believes may increase the risk of the subject or interfere with the results of the test;

Ages: 2 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-12-16 (Actual); Primary Completion 2021-12-16 (Estimated); Study Completion 2022-02-16 (Estimated)

PRIMARY OUTCOMES:
Safety: Incidence and severity of adverse events | First 1 month post CAR-T cells infusion
  To evaluate the possible adverse events occurred within first one month after CAR-γδT infusion, including the incidence and severity of symptoms such as cytokine release syndrome and neurotoxicity
Efficacy: Remission Rate | 3 months post CAR-T cells infusion
  Remission Rate including complete remission(CR)、CR with incomplete blood count recovery(CRi)、No remission(NR)

SECONDARY OUTCOMES:
duration of response (DOR) | 24 months post CAR-T cells infusion
  duration of response (DOR)
Efficacy: progression-free survival (PFS) | 24 months post CAR-T cells infusion
  progression-free survival (PFS) time
CAR-T proliferation | 3 months post CAR-T cells infusion
  the copy number of CAR- γδT cells in the genomes of PBMC by qPCR method
Cytokine release | First 1 month post CAR-T cells infusion
  Cytokine( IL-6,IL-10,IFN-γ,TNF-α ) concentration (pg/mL) by flow cytometry method

CONTACTS AND LOCATIONS:
Overall Officials: Peihua MD Lu, PhD, Principal Investigator — Hebei Yanda Ludaopei Hospital
Locations (1):
- Hebei yanda Ludaopei Hospital, Yanda, Hebei, China